CLINICAL TRIAL: NCT06980272
Title: A Randomized Controlled, Multi-center Phase III Clinical Trial of SSGJ-707 Versus Pembrolizumab as First-line Treatment for PD-L1-Positive Locally-Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: SSGJ-707 in Advanced Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-707-NSCLC-III-01
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-05

CONDITIONS: Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSGJ-707 (Experimental): Subjects receive SSGJ-707 monotherapy intravenously (IV), selected dose.
  Interventions: Drug: SSGJ-707
- Pembrolizumab (Active Comparator): Subjects receive Pembrolizumab monotherapy intravenously (IV), 200mg q3w.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: SSGJ-707 — Subjects receive SSGJ-707 intravenously.
  Arms: SSGJ-707
Drug: Pembrolizumab — Subjects receive Pembrolizumab intravenously.
  Arms: Pembrolizumab

SUMMARY:
This trial is a Phase III study. All patients are stage IIIB/C (unsuitable for radical therapy) or IV non-small cell lung cancer(NSCLC), Eastern Cooperative Oncology Group (ECOG) performance status 0-1. The purpose of this study is to evaluate the efficacy and safety of SSGJ-707 comparing Pembrolizumab in subjects with advanced NSCLC whose tumors have a programmed cell death-ligand 1 (PD-L1) Tumor Proportion Score (TPS) greater than or equal to 1%.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study voluntarily, agree to comply with and complete all study procedures, and sign the Informed Consent Form (ICF).
2. At least 18 years of age at the time of signing the ICF, regardless of gender.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
4. Life expectancy of at least 12 weeks.
5. Histologically or cytologically confirmed locally advanced (Stage IIIB/IIIC) or metastatic (Stage IV) non-small cell lung cancer (NSCLC).
6. No prior systemic anti-tumor treatment for locally advanced or metastatic NSCLC.
7. At least one measurable tumor lesion as a target lesion according to RECIST v1.1 criteria.

Exclusion Criteria:

1. Presence of small cell carcinoma components in histological pathology.
2. Presence of EGFR-sensitive mutations or ALK fusion-positive NSCLC.
3. Known BRAF V600E mutation, MET exon 14 skipping mutation, NTRK fusion, RET fusion, or ROS1 fusion-positive NSCLC.
4. Presence of brainstem, leptomeningeal, spinal cord metastasis or compression.
5. Unresolved toxicity from prior anti-tumor treatment, defined as toxicity not returning to NCI CTCAE Version 5.0 Grade 0 or 1.
6. History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
7. History of immunodeficiency; positive for HIV antibodies;
8. Known active tuberculosis (TB);
9. Known history of severe allergy to any component of the investigational drug, or history of severe allergic reactions to chimeric or humanized antibodies.
10. Pregnant or breastfeeding women.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by IRRC per RECIST v1.1 | Up to 2 approximately years
  Progression-free survival (PFS) is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the blinded IRRC or death due to any cause (whichever occurs first).

SECONDARY OUTCOMES:
OS | Up to 2 approximately years
  Overall Survival (OS) is defined as the time from the start of treatment with SSGJ-707 until death due to any cause.
ORR assessed by IRRC per RECIST v1.1 | Up to 2 approximately years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1.
DoR assessed by IRRC per RECIST v1.1 | Up to 2 approximately years
  Duration of response (DoR) assessed according to RECIST v1.1.
DCR assessed by IRRC per RECIST v1.1 | Up to 2 approximately years
  Disease control rate (DCR) assessed according to RECIST v1.1.
TTR assessed by IRRC per RECIST v1.1 | Up to 2 approximately years
  Time to response (TTR) is defined as the time to response base on RECIST v1.1.
PFS assessed by investigator per RECIST v1.1 | Up to 2 approximately years
  Progression-free survival (PFS) is defined as the time from the date of randomization till the first documentation of disease progression assessed by the investigator or death due to any cause (whichever occurs first).
ORR assessed by the investigator per RECIST v1.1 | Up to 2 approximately years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1.
DoR assessed by the investigator per RECIST v1.1 | Up to 2 approximately years
  Duration of response (DoR) assessed according to RECIST v1.1.
DCR assessed by the investigator per RECIST v1.1 | Up to 2 approximately years
  Disease control rate (DCR) assessed according to RECIST v1.1.
TTR assessed by the investigator per RECIST v1.1 | Up to 2 approximately years
  Time to response (TTR) is defined as the time to response base on RECIST v1.1.
AE | Up to 2 approximately years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
ADA | Up to 2 approximately years
  Number of subjects with detectable anti-drug antibodies (ADA).
PD-L1 expression | Up to 2 approximately years
  The correlationship between PD-L1 expression and SSGJ-707 anti-tumor activity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Shanghai East Hospital, Shanghai, China